CLINICAL TRIAL: NCT05847491
Title: Latent Tuberculosis in Healthcare Workers - the Reality of a Portuguese Tertiary Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Hospitalar do Oeste (Other)
Responsible Party: Sponsor
Other Study IDs: LTBCHO23
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Tuberculosis
Keywords: Latent Tuberculosis; Healthcare workers; IGRA
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthcare workers: Clinical evaluation, chest x-ray and Interferon-γ release assay (IGRA). Immunocompromised patients will be submitted to a tuberculin skin test.
  The patients will be evaluated in two or more separate appointments. In the first appointment, patients will be submitted to clinical evaluation and exam request. In the second appointment the results will be evaluated.
  Interventions: Diagnostic Test: IGRA/Tuberculin skin test

INTERVENTIONS:
Diagnostic Test: IGRA/Tuberculin skin test — All patients will receive:
  * Clinical evaluation;
  * Chest x-ray.
  * IGRA (or tuberculin skin test if immunocompromised)
  * Therapeutic proposal if eligible

SUMMARY:
Prospective, descriptive study to assess latent tuberculosis infection (LTBI) among healthcare worker (HCW) in a tertiary hospital in a low-risk area.

DETAILED DESCRIPTION:
identiﬁcation and treatment of LTBI can substantially reduce the risk of development of disease and are important TB control strategies, especially in settings with a low tuberculosis (TB) incidence, where reactivation of LTBI often accounts for the majority of non-imported TB disease treatment of LTBI can substantially reduce the risk of development of disease.

In Portugal the real prevalence of LTBI in low-risk HCWs has not been evaluated since they are not included in the periodic screening programs. It is important to diagnose TB infections in HCWs to prevent nosocomial transmission, particularly among immunocompromised patients.

The risk for transmission varies by setting, occupational group, local prevalence of TB, patient population, and effectiveness of TB infection control measures.

Prevention of active TB disease by treatment of LTBI is a critical component for public health.

Tuberculin skin test (TST) is used worldwide to diagnose LTBI, whereas interferon-γ release assay (IGRA) are used in some countries according to their national TB programs. IGRA offers a potential method of serial testing to diagnose LTBI in HCWs, and it has better specificity than that of TST in one-time screening.

Study participants should be identified and contacted by occupational health service. In association, study information should be disseminated through posters and institutional email.

ELIGIBILITY:
Inclusion Criteria:

* All HCW from our hospital with risk of exposure, working in our hospital for at least 3 consecutive months
* Acceptance to participate and signed informed consent form

Exclusion Criteria:

* History of previous tuberculosis
* Active Tuberculosis
* Refusal to sign the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical staff, nurses, laboratory, cardiopulmonary and radiology technician, operational staff from our hospital working for 3 or more months.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of latent tuberculosis diagnosis in healthcare workers | 1 year
  Patients with positive IGRA/tuberculin test screening and without clinical or radiological features of active Tuberculosis

SECONDARY OUTCOMES:
Treatment acceptance for latent tuberculosis | 1 year
  Number of positive screening participants who accept and start treatment
Treatment completion | 1 year
  Number of patients who finished treatment

OTHER OUTCOMES:
Treatment discontinuation | 1 year
  Number of patients who did not complete treatment

CONTACTS AND LOCATIONS:
Overall Officials: Carina Rolo Silvestre, MD, MSc, Principal Investigator — Centro Hospitalar do Oeste
Locations (1):
- Centro Hospitalar do Oeste - Torres Vedras, Torres Vedras, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication.
Supporting Information: Study Protocol, ICF
Time Frame: After publication.
Access Criteria: By request to the authors.

REFERENCES:
- [Background] Adams S, Ehrlich R, Baatjies R, van Zyl-Smit RN, Said-Hartley Q, Dawson R, Dheda K. Incidence of occupational latent tuberculosis infection in South African healthcare workers. Eur Respir J. 2015 May;45(5):1364-73. doi: 10.1183/09031936.00138414. Epub 2015 Feb 19. PMID 25700382
- [Background] Almufty HB, Abdulrahman IS, Merza MA. Latent Tuberculosis Infection among Healthcare Workers in Duhok Province: From Screening to Prophylactic Treatment. Trop Med Infect Dis. 2019 May 23;4(2):85. doi: 10.3390/tropicalmed4020085. PMID 31126022
- [Background] Apriani L, McAllister S, Sharples K, Alisjahbana B, Ruslami R, Hill PC, Menzies D. Latent tuberculosis infection in healthcare workers in low- and middle-income countries: an updated systematic review. Eur Respir J. 2019 Apr 18;53(4):1801789. doi: 10.1183/13993003.01789-2018. Print 2019 Apr. PMID 30792341
- [Background] Chen B, Gu H, Wang X, Wang F, Peng Y, Ge E, Upshur R, Dai R, Wei X, Jiang J. Prevalence and determinants of latent tuberculosis infection among frontline tuberculosis healthcare workers in southeastern China: A multilevel analysis by individuals and health facilities. Int J Infect Dis. 2019 Feb;79:26-33. doi: 10.1016/j.ijid.2018.11.010. Epub 2018 Nov 22. PMID 30471404
- [Background] Costa JC, Silva R, Ferreira J, Nienhaus A. Active tuberculosis among health care workers in Portugal. J Bras Pneumol. 2011 Sep-Oct;37(5):636-45. doi: 10.1590/s1806-37132011000500011. English, Portuguese. PMID 22042396
- [Background] Park Y, Kim SY, Kim JW, Park MS, Kim YS, Chang J, Kang YA. Serial testing of healthcare workers for latent tuberculosis infection and long-term follow up for development of active tuberculosis. PLoS One. 2018 Sep 20;13(9):e0204035. doi: 10.1371/journal.pone.0204035. eCollection 2018. PMID 30235272